CLINICAL TRIAL: NCT05380063
Title: Ticagrelor-based De-escalation of Dual Antiplatelet Therapy After Coronary Artery Bypass Grafting in Patients Without Acute Coronary Syndrome
Brief Title: Ticagrelor-based De-escalation of Dual Antiplatelet Therapy After Coronary Artery Bypass Grafting
Acronym: TOP-CABG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Shengshou Hu, Professor, China National Center for Cardiovascular Diseases
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-ZX100
Record Dates: First submitted 2022-05-13; First posted 2022-05-18 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-07

CONDITIONS: Coronary Artery Disease; Coronary Artery Bypass Grafting; Dual Antiplatelet Therapy; Bleeding; Myocardial Infarction; Myocardial Ischemia; Angina Pectoris
Keywords: Coronary Artery Bypass Grafting; Ticagrelor; Aspirin; Dual Antiplatelet Therapy; De-escalated Dual Antiplatelet Therapy; Great Saphenous Vein; Bleeding
MeSH Terms: conditions — Coronary Artery Disease; Hemorrhage; Myocardial Infarction; Myocardial Ischemia; Angina Pectoris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dual Antiplatelet Therapy (DAPT) (Active Comparator): DAPT with ticagrelor (90mg twice daily) + aspirin (100 mg once daily) for 1 year after CABG.
  Interventions: Drug: Dual Antiplatelet Therapy
- De-escalated Dual Antiplatelet Therapy (De-DAPT) (Experimental): De-DAPT referred to ticagrelor (90mg twice daily) + aspirin (100 mg once daily) during first 3 months post CABG, then switch to aspirin (100 mg once daily) + placebo (twice daily) for 9 months.
  Interventions: Drug: De-escalated Dual Antiplatelet Therapy

INTERVENTIONS:
Drug: De-escalated Dual Antiplatelet Therapy — ticagrelor (90mg twice daily) + aspirin (100 mg once daily) during first 3 months post CABG, then switching to aspirin (100 mg once daily) + placebo (twice daily) for 9 months.
  Other Names: De-escalation
  Arms: De-escalated Dual Antiplatelet Therapy (De-DAPT)
Drug: Dual Antiplatelet Therapy — Ticagrelor (90mg twice daily) + aspirin (100 mg once daily) for 1 year post CABG.
  Arms: Dual Antiplatelet Therapy (DAPT)

SUMMARY:
Ticagrelor-based De-escalation of Dual Antiplatelet Therapy After Coronary Artery Bypass Grafting trial (TOP-CABG trial) is a multicenter, randomized, double-blind, non-inferiority, parallel controlled trial. The aim of TOP-CABG is to investigate whether de-escalated dual antiplatelet therapy (De-DAPT) is non-inferior to dual antiplatelet therapy (DAPT) in efficacy on inhibiting great saphenous vein (SVG) graft occlusion and is superior in reducing bleeding events in patients accepting coronary artery bypassing grafting.

DETAILED DESCRIPTION:
After informed consent, at least 10 centers and 2,300 eligible admissions will be recruited. Eligible patients would be randomized (1:1) in double-blind manner (patients and treating physicians) to dual antiplatelet therapy (DAPT) group (ticagrelor 90mg bid and aspirin 100 mg qd for 12 month) and de-escalated DAPT (De-DAPT) group (90mg bid and aspirin 100 mg qd for first 3 months, and then aspirin 100 mg qd and placebo for 9 months).

ELIGIBILITY:
Inclusion criteria

1. Patients 18-80 of age. 2. Patients undergo planned CABG for the first time with ≥1 SVGs 3. Patients with written informed consent. Exclusion criteria

1. Concomitant valve (excluding aortic bioprosthesis), aorta, or rhythm surgery during the same session.
2. Patients undergo emergency CABG.
3. Patients with single coronary artery disease.
4. Patients with cardiogenic shock and hemodynamic instability.
5. Patients with sick sinus syndrome, 2nd or 3rd atrioventricular block.
6. Patients with contraindications for coronary computed tomography angiography or coronary angiography (eg. contrast allergy).
7. Use of other antiplatelet drugs than aspirin or ticagrelor (clopidogrel, prasugrel, etc) and unable to discontinue this medication after CABG, in the treating physician's or the investigator's opinion.
8. Patients who take oral anticoagulants before CABG and have to use anticoagulants after surgery.
9. Contraindication for the use of ticagrelor or aspirin (ie. history of bleeding diathesis within 3 months prior presentation, severe gastrointestinal bleeding within 1year prior presentation, peptic ulcer without gastrointestinal bleeding in past 3 years or history of intracranial hemorrhage, allergy, severe gastrointestinal reaction caused by aspirin).
10. Placement of a drug-eluting stent in a coronary or cerebral artery within 6 months of CABG or placement of a bare-metal stent in a coronary or cerebral artery within 1 month of CABG
11. Thrombocytopenia before CABG (< 100 x 109/L).
12. patients with severe renal function impairment requiring dialysis or active liver disease, including patients with unexplained persistent elevated transaminase or any transaminase more than 3 times the normal limit.
13. Use of strong inhibitors of CYP3A4
14. Patients who have to use methotrexate and ibuprofen.
15. Patients with active malignant tumors with increase in bleeding risk in the investigator's opinion
16. Pregnant patients, patients who have given birth within the past 90 days, or who are breastfeeding.
17. Premenopausal women who do not take adequate contraception. Adequate contraception refers to the adoption of at least two reliable methods of contraception, one of which must be a barrier method of contraception.
18. CABG volume of the surgeon less than 50.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2300 (Actual)
Dates: Start 2023-02-14 (Actual); Primary Completion 2025-07-08 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
100% great saphenous vein (SVG) grafts occlusions | During 0-day to 1-year after CABG
  100% SVG During 0-day to 1-year after CABG (Fitz Gibbon grade O). SVG grafts were assessed by multislice computed tomographic angiography or coronary angiography and interpreted by an independent Image Data Review Centre blinded to treatment allocation
Bleeding events | During 0-day to 1-year after CABG
  Bleeding events as defined by the BARC classification ≥ 2 at 1 year after CABG.

SECONDARY OUTCOMES:
SVG Failure | During 0-day to 1-year after CABG
  a composite of SVG occlusion in any SVG as defined above, SVG revascularization, myocardial infarction in myocardial territory supplied by an SVG, or sudden death, as defined by the American College of Cardiology and American Heart Association and judged by an independent Clinical Endpoint Committee blinded to treatment allocation
Graft stenosis and occlusion | During 0-day to 1-year after CABG
  Significant (≥70%) venous or arterial graft stenosis and any (venous or arterial) graft occlusion
MACCE episodes | Within 1-year after CABG
  MACCE episodes within 1-year after CABG (composite of cardiovascular death, nonfatal myocardial infarction, nonfatal stroke or revascularization), as defined by the American College of Cardiology and American Heart Association and judged by an independent Clinical Endpoint Committee blinded to treatment allocation

OTHER OUTCOMES:
Subgroup analysis 1 for primary outcome | 1 year
  Age (<65 years, ≥65 years)
Subgroup analysis 2 for primary outcome | 1 year
  Sex (male, female)
Subgroup analysis 3 for primary outcome | 1 year
  Body mass index (<25 kg/m2, ≥25 kg/m2)
Subgroup analysis 4 for primary outcome | 1 year
  Acute Coronary Syndrome (yes, no)
Subgroup analysis 5 for primary outcome | 1 year
  Hypertension (yes, no)
Subgroup analysis 6 for primary outcome | 1 year
  Diabetes (yes, no)
Subgroup analysis 7 for primary outcome | 1 year
  Dyslipidemia (yes, no)
Subgroup analysis 8 for primary outcome | 1 year
  Prior myocardial infarction (yes, no)
Subgroup analysis 9 for primary outcome | 1 year
  Current smoker (yes, no)
Subgroup analysis 10 for primary outcome | 1 year
  Left ventricular ejection fraction (<50%, ≥50%)
Subgroup analysis 11 for primary outcome | 1 year
  eGFR (<60/ml/min/1.75m2, ≥60/ml/min/1.75m2)
Subgroup analysis 12 for primary outcome | 1 year
  Statin (yes, no)
Subgroup analysis 13 for primary outcome | 1 year
  Beta-blocker (yes, no)
Subgroup analysis 14 for primary outcome | 1 year
  RASi (yes, no)
Subgroup analysis 15 for primary outcome | 1 year
  Off-pump (yes, no)
Subgroup analysis 16 for primary outcome | 1 year
  Grafts (<3 , ≥3)
Subgroup analysis 17 for primary outcome | 1 year
  Syntax score(≤22, 23-32 , ≥33)

CONTACTS AND LOCATIONS:
Overall Officials: Shengshou Hu, MD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital; Xin Yuan, PhD, Study Chair — Chinese Academy of Medical Sciences, Fuwai Hospital; Qing Chu, PhD, Study Director — Chinese Academy of Medical Sciences, Fuwai Hospital; Kai Chen, Study Director — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yuan X, Chu Q, Chen K, Wang Y, Zhang L, Zheng Y, Hu S. Multicentre, randomised, double-blind, parallel controlled trial to investigate timing of platelet inhibition after coronary artery bypass grafting: TOP-CABG trial study. BMJ Open. 2023 Jun 29;13(6):e070823. doi: 10.1136/bmjopen-2022-070823. PMID 37385747